CLINICAL TRIAL: NCT07058116
Title: Accelerator-based Boron Neutron Capture Therapy (BNCT) in the Treatment of Locally Recurrent Head and Neck Carcinoma: A Phase I Study.
Brief Title: Accelerator-based BNCT (Boron Neutron Capture Therapy) for Head and Neck Carcinoma.
Acronym: BNCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neutron Therapeutics, LLC (Industry)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-BNCT-01-2024; 2024-515036-71-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Carcinoma
Keywords: L-Boronophenylalanine; BNCT; Boron Neutron Capture Therapy; Head and Neck Carcinoma; Neutron Therapeutics; Helsinki University Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group - Dose escalation study (Experimental): Two BNCT trial treatments are scheduled to be administered to each study subject with a 4-week time interval between the 2 trial treatments (a range from 3.0 to 6.0 weeks is allowed for the interval). Neutron irradiations are given at the Helsinki University Hospital BNCT facility (Helsinki, Finland) using the nuBeam Suite. The nuBeam Treatment Delivery System within the nuBeam Suite delivers a neutron beam that has suitable energy and flux for clinical BNCT.
  The Instructions for Use/User Guide(s) containing the detailed instructions for using the system will be followed for the delivery of neutron irradiation for each BNCT trial treatment.
  The basic steps for the irradiation procedure are:
  1. Neutron source preparation/calibration
  2. CT imaging of the target region
  3. Positioning of the study subject
  4. Irradiation to the planned trial treatment dose
  5. Close-out/Shutdown Each BNCT trial treatment will be carried out according to the trial treatment plan.
  Interventions: Drug: L-Boronophenylalanine intravenous administration

INTERVENTIONS:
Drug: L-Boronophenylalanine intravenous administration — L-BPA will be complexed with fructose to form L-BPA-fructose (L-BPA-F) to increase solubility, and 400 mg/kg of L-BFA as complexed with fructose (L-BPA-F) will then be administered intravenously at a concentration of L-BPA 30 g/L over 2 hours before neutron irradiation.
  Other Names: Neutron Irradiation

SUMMARY:
This phase I study of an accelerator-based boron neutron capture therapy (BNCT) in the treatment of locally recurrent head and neck carcinoma, is sponsored by HUS, Haartmaninkatu 4, Helsinki, Finland and Neutron Therapeutics Finland OY, Kanavaranta 9 FIN-00290 Helsinki.

The indication is for patients with head and neck carcinoma that has recurred locally after conventional radiation therapy.

The primary objective is to demonstrate the safety of accelerator-based neutron radiation using the nuBeam Suite in delivering BNCT.

The secondary objective is the ability to deliver the planned radiation dose to the target site and the ability to plan the trial treatment using the trial treatment planning software, position and target the tumor site using the robotic table in conjunction with the CT scanner and calculate the required radiation dose for each planned BNCT trial treatment.

To establish these objectives, the following parameters will be controlled:

* Objective response rate
* Duration of response.
* The clinical benefit rate (includes complete response, partial response, and stabilized disease for a minimum of 8 weeks since the date of the first BNCT).
* Locoregional recurrence-free survival.
* Progression-free survival.
* Overall survival.
* Quality of life.

The maximum sample size is 10 study subjects evaluable for safety.

The study does not involve randomization.

Regarding the target population, the study subjects must fulfill each of the inclusion criteria:

1. Patient has provided a written informed consent as approved by the EC prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. ≥ 18 years of age at the time of enrollment.
3. Histologically confirmed head and neck carcinoma.
4. Inoperable cancer, prior surgery may or may not have been done.
5. Prior radiotherapy or chemoradiotherapy has been given.
6. Anticipated life expectancy of at least 6 months

Patients who fulfill any of the following criteria will be excluded:

1. Presence of distant metastases.
2. World Health Organization (WHO) performance status > 2
3. Concurrent uncontrolled localized cancer other than head and neck carcinoma or overtly metastatic cancer.
4. The patient has access to a non-experimental, effective treatment option and is a suitable candidate for such therapy.
5. Concomitant chemotherapy.
6. Concurrent experimental therapy or participation in a trial with an experimental therapy within 3 months prior to study inclusion.
7. Less than 3 months since prior radiation therapy.
8. Major surgery within 4 weeks prior to study inclusion.
9. Unremovable metal implants present in the head and neck region that will interfere with CT/MRI-based dose-planning.
10. Known sensitivity to the study drug.
11. One or more of the following:

    * Blood hemoglobin < 100 g/L, neutrophils < 1.5 x 109/L, platelet count < 120 x 109/L
    * Serum/plasma creatinine > 1.5 x Upper Limit of Normal (ULN)
    * Serum bilirubin 2.0 > ULN
    * Serum ALT and/or AST > 2.0 x ULN
    * Serum alkaline phosphatase > 2.5 x ULN
12. Serious uncontrolled infection or other serious uncontrolled concomitant disease.
13. Collagen vascular disease or a disease that is considered to increase radiosensitivity of normal tissues to radiation (e.g., ataxia-telangiectasia)
14. Patient is unwilling or unable to comply with the CIP required follow-up visits for the duration of the study.
15. Untreated or severe treated congestive heart failure, cardiac pacemaker, or renal failure.
16. Restlessness or inability to lie in a cast for about 30 minutes.
17. Clinical follow-up after therapy cannot be arranged or the patient is not willing to participate in the follow-up.
18. Known pregnancy, breastfeeding, or planning of pregnancy; for women of childbearing potential, a negative pregnancy test must be obtained prior to enrollment.
19. The patient is not able to understand the nature of the study and trial treatment options.
20. Phenylketonuria
21. Fructose intolerance.

There is one investigational device included as part of this study. The nuBeam Suite has two main components, the Treatment Delivery System and the nuBeam Dose Engine.

The study drug included in this study is L-boronophenylalanine fructose (L-BPA Fructose)

DETAILED DESCRIPTION:
CLINICAL STUDY BACKGROUND AND RATIONALE

Disease Background and Unmet Clinical Need Head and neck carcinoma accounts for about 5% of all cancers and is the sixth most common type of cancer in humans. More than 650,000 new cases are detected annually worldwide, leading to more than 350,000 deaths. Head and neck carcinoma comprise carcinomas located in the oral cavity, the nasopharynx, the oropharynx, the hypopharynx, the larynx, the paranasal sinuses, and the salivary glands. Some carcinomas are related to smoking or alcohol abuse, but an increasing proportion of oropharynx and tonsil carcinomas, in particular, are related to human papilloma virus (HPV) infection. Cancer HPV status is often determined with immunohistochemistry from the cancerous tissue by demonstrating positive immunostaining for p16, an inhibitor of cyclin-dependent kinases 4 and 6. p16 is upregulated in HPV-infected tissues with inactivated retinoblastoma protein. Nasopharynx carcinomas are also frequently associated with oncogenic viruses.

Most patients with head and neck carcinomas have squamous cell carcinoma of the head and neck (HNSCC), and present with locally advanced stage disease. Several factors need to be considered when selecting for the trial treatment, including the primary tumor size and location, presence of metastases, the histological type and histological features of cancer, depth of cancer invasion, patient performance status and comorbidities, and whether cancer is HPV infection related or not. In general, early carcinomas may be treated with a single treatment modality, whereas advanced carcinomas require a multimodality approach for achieving optimal outcomes. Surgery and radiation therapy are the mainstay of locoregional treatment. Radiation therapy is often given concomitantly with certain chemotherapy agents, notably platin salts, to improve efficacy. Precision radiotherapy, such as intensity modulated radiotherapy (IMRT), reduces some adverse effects including xerostomia, and improves locoregional cancer control. New radiotherapy techniques such stereotactic ablative radiotherapy (SABR) and proton therapy are under active evaluation.

Although substantial advances have been made in the treatment of HNSCC, still 20% to 50% of the patients treated with chemoradiotherapy for unresectable HNSCC have locoregional cancer recurrence. Distant metastases are not uncommon, and survival outcomes remain relatively poor also in locally advanced disease. The overall long-term survival of patients with head and neck carcinoma is about 50% but varies greatly depending on factors such as tumor size, site, and the histological type.

Locoregionally recurrent HNSCC is usually treated with surgery, radiation therapy, and/or systemic therapy. The preferred option for operable patients is salvage surgery, which leads to 5-year survival up to 40%. Many recurrent cancers are, however, considered inoperable, or surgery is anticipated to lead to substantial morbidity. Reirradiation is an option for selected. The reported survival outcomes vary depending on patient selection and the techniques used with 2-year overall survival ranging from 10% to 35%. Cumulative doses greater than 60 Gy are usually recommended for reirradiation despite the relative high frequency of severe adverse events associated with such treatments. In recent years, a growing body of literature has reported on the safety and feasibility of hypofractionated radiotherapy for tumors of the head and neck. Most of these series include patients with recurrent, unresectable head and neck carcinomas who had been previously irradiated. These studies have found promising overall response rates up to 80% and 1-year local control rates in the range of 50% Chemotherapy with or without an agent targeted for the epidermal growth factor receptor (EGFR, HER1) has moderate efficacy, but is not considered curative if administered alone. Some patients respond to immune therapy obtaining clinically meaningful objective responses.

In sum, although the treatment of locoregionally recurred head and neck carcinoma has evolved substantially during the recent years, the disease is frequent ultimately lethal, and the current therapies may be associated with substantial morbidity. Therefore, there is a clinical need to improve the treatment results in locally recurred head and neck carcinoma, and novel approaches are urgently needed.

Boron Neutron Capture Therapy (BNCT)

BNCT has several potential advantages compared to conventional radiation therapy. First, BNCT has the capability of treating tumors that are highly infiltrating into sensitive tissues where surgery with effective margins would be impossible or mutilating. In addition to the potentially increased effectiveness, this approach as delivered by the nuBeam System is anticipated to provide quality of life benefits due to the reduced side-effects, simplified procedure and reduced cosmetic consequences of the trial treatment as seen in research.

The high-LET (Linear Energy Transfer) radiation produced by BNCT also conveys several advantages. It produces double-strand DNA breaks and should do so even in hypoxic conditions where conventional radiation therapy loses effectiveness. The mechanism of action of high-LET radiation has also been shown to be effective in treating radio-resistant cancers. High-LET in combination with BNCT's ability to effectively spare healthy tissue also allows trial treatments to be carried out in only one or two fractions, which leads to improved patient quality of life as well as the potential for cost reduction when compared to conventional courses of radiation therapy, typically requiring as many as 35 fractions.

BNCT is based on the neutron capture and fission reactions that occur when non-radioactive boron (10B) is irradiated with neutrons of low (thermal) energy (0.025 eV). This causes boron nuclear decay, which yields high linear energy transfer (LET) α particles (4He) and recoiling lithium (7Li) nuclei. Alternatively, to improve neutron tissue penetration, epithermal (10 keV) neutrons that become thermalized (lost energy) in tissue may be used. Since α and 7Li have only a short range in tissue (5 to 9 µm) and they produce dense ionization along their tracks, most radiation effect is local and occurs within the cells that contain boron. The success of BNCT depends upon a selective uptake of sufficient amounts of 10B into cancer cells compared with normal tissues (approximately 20 to 50 µg/g; 109 atoms per cancer cell).

Selective accumulation of boron into cancerous tissue can be achieved using a boron carrier compound that is preferentially taken up by cancer. The most frequently used agents to deliver boron are a derivative of the amino acid phenylalanine, L-boronophenylalanine (L-BPA), sodium borocaptate (BSH), or their combination. After administration of the boron carrier compound (usually using an intravenous infusion), the tumor is irradiated with neutrons.

Until recently, the source of the neutrons needed for BNCT has been a nuclear reactor. This has been a limitation, since nuclear reactors are an expensive neutron source, they are often located at remote sites and are only infrequently available for medical use, and the beam obtained from nuclear reactors requires moderation to obtain neutrons with a suitable flux and energy for BNCT. At present, nuclear reactor-based BNCT is only rarely available for clinical purposes. However, neutron beams with characteristics suitable for BNCT can now be obtained with particle accelerators. A few companies, including three Japanese companies, Hitachi, Sumitomo Heavy Industries, and Mitsubishi Heavy Industry Co., and one American company, Neutron Therapeutics, have built an accelerator neutron source for BNCT. Phase I/II clinical BNCT trials, based on accelerator technology, have been conducted in Japan with promising antitumor effects and good safety, and are planned to be initiated in Finland with this clinical investigation.

Several hundreds of patients have been treated with BNCT using neutrons obtained from a nuclear facility and with L-BPA and/or BSH as the boron carrier. Most patients have had either malignant glioma, head and neck carcinoma, melanoma, or meningioma, but a few patients with other types of tumors have also been treated. In general, BNCT has been relatively well tolerated even in patients who have already been treated with conventional radiation therapy or chemoradiation, the most frequent adverse events being similar to those associated with conventional radiation therapy. The adverse events related to L-BPA and BSH have been few, and both agents thus seem generally well tolerated boron carriers when administered intravenously at the dosages used in clinical trials.

The median survival time of patients with newly diagnosed glioblastoma has been approximately 1 year when they have been treated with surgery and BNCT. This duration is approximately similar to that obtained with surgery followed by conventional radiotherapy when administered without temozolomide. L-BPA-mediated BNCT can be administered also to patients who have glioblastoma that has recurred after surgery and conventional radiotherapy. Such patients survived for a median of about 7 months, and BNCT was generally well tolerated.

Most patients with locally recurred, inoperable head and neck cancer treated in nonrandomized Phase I/II trials with BNCT respond to BNCT. The response rate was about 70 % (range, from 58% to 90%) with a complete response (CR) achieved in 55%. The most common adverse events were mucositis, oral pain, and fatigue. As with other therapies, recurrence is frequent in this patient population. In a trial carried out in Finland the 2-year locoregional recurrence-free survival was 27%, 2-year progression-free survival 20%, and 2-year overall survival 30%. In sum, these data suggest that BNCT is effective and moderately well tolerated in the treatment of locally recurrent, inoperable head and neck cancer leading to relatively high response rates.

Limited data suggest that BNCT can be combined with conventional radiotherapy and with some systemic agents in the treatment of head and neck cancer, but in the absence of clinical trials such an approach remains experimental. Besides head and neck carcinoma, BNCT appears effective also in the treatment of some other human tumor types, such as melanomas of the extremities, and aggressive meningiomas.

Rationale of the Clinical Study Locally recurred head and neck carcinoma poses a substantial therapeutic challenge. Most such cancers eventually progress regardless of the type of therapy, and the majority of cancer progressions eventually lead to death resulting from either local cancer progression, distant metastases, or both. There is a clear unmet need for more effective treatments and for novel treatment options.

As discussed above, L-BPA-mediated BNCT has resulted in promising clinical results in prior clinical studies using reactor-based neutron sources in Finland, Japan, Taiwan and elsewhere. Recent technical innovations have led to the development of proton accelerator-based neutron sources that are suitable for BNCT and can be installed in hospital environments. Such neutron sources can be designed specifically for hospital use, with a focus on reliability and simplicity of operation. Their performance characteristics can be tailored to closely mirror the proven FiR-1 reactor BNCT installation, with similar radiation quality and moderately improved epithermal neutron flux. Accelerator-based systems can be outfitted with automated patient imaging and positioning features to allow for improved targeting of radiation to the tumor and cost-effective treatment of a large number of patients. Next-generation BNCT devices can also be linked to modern treatment planning software platforms, enabling optimized planning of the radiation fields to minimize collateral dose and reduce complication rates.

Taken together, there is a strong rationale to study the safety, performance and efficacy of accelerator-based BNCT with infused L-BPA in the trial treatment of locally recurrent head and neck carcinoma.

The proposed BNCT trial treatment comprises the nuBeam Suite: a set of devices for administering BNCT including an investigational Therapeutic Neutron Source, and L-boronophenylalanine, a boron carrier compound. Both components are required in order to administer BNCT: the device to deliver epithermal neutrons to the target region and the drug to concentrate the neutron-absorbing boron isotope to the cancer cells.

This study is an exploratory clinical investigation according to ISO/FDIS 14155:2020(E) - Annex I. Results from this study will be used to guide development and refinement of accelerator-based boron neutron capture therapy.

The nuBeam Suite is a comprehensive tool for administering neutron capture therapy (NCT) from planning through image guided delivery of the therapeutic neutron radiation. It is composed of two distinct devices: the Treatment Delivery System (TDS) and the NCT Planning System.

The nuBeam TDS has two main components:

1. Therapeutic Neutron Source (TNS), with integrated Treatment Control System and Patient Position Verification System (PPVS)
2. Patient Positioning and Imaging System (PIPS)

   * Therapeutic Neutron Source, a product of Neutron Therapeutics (Finland/USA) Therapeutic Neutron Source (TNS) is the main non-CE Marked investigational device in this clinical study. The TNS creates the neutron beam, monitors the fluence of neutrons delivered, and controls the irradiation including loading and performing of an irradiation plan. The device does not contain any sterile or single use components.
   * Patient Imaging and Positioning System, a product of BEC GmbH (Germany)

The Patient Positioning and Imaging System (PIPS) within the nuBeam Suite consists of the BEC Exacure System, which has two main modules: Examove and Exaview. Examove is based on an industrial six-axis robot from KUKA, programmed and outfitted for use in a medical environment. It is ceiling-mounted on a 7th axis linear rail, which provides the necessary accuracy and versatility to conduct the desired positioning and imaging operations. This axis also allows the base of the robot to be positioned well away from the neutron beam, reducing neutron scatter back to the patient. Exaview integrates the robot with a rail mounted Siemens Healthineers Somatom Confidence® CT scanner (a CE Marked device) to take in-room CT images to compare with the planning images for precise patient positioning. Exacure was first developed and deployed for the MedAustron proton/carbon ion center in Austria and has undergone extensive neutron sensitivity testing.

The additional features that were added to the BEC Exacure System for the nuBeam Suite are part of the CE mark.

The features added include:

* Suitable components and material selection (e.g. avoidance of aluminum)
* Component positioning (e.g. outsourced robot controller components)
* Shielding of the linear axis, robot, tracking camera

  * The Patient Position Verification System, a product of Cosylab (Slovenia)/Neutron Therapeutics (Finland/USA) The Patient Position Verification System (PPVS) within the nuBeam Suite consists of the Cosylab ImageOne PPVS. This product uses the CT images from the irradiation plan and compares them with the in-room CT images acquired by the PIPS. The system then aligns the two images providing a six degree of freedom correction vector to the Cosylab TreatmentOne Treatment Control System (TCS) with submillimeter accuracy.

The NCT Planning System also consists of two components:

* RayStation Treatment Planning System
* nuBeam Dose Engine
* RayStation NCT Treatment Planning System, a product of RaySearch Laboratories (Sweden) RayStation® Treatment Planning software is widely used for radiation therapy. RaySearch has developed a new version called RayStation-NCT software which is capable of NCT planning. This functionality is enabled via a special license activated in the nuBeam Suite. RayStation is CE marked after each version release and Raystation-NCT may be CE Marked prior to commencement of the clinical investigation.
* nuBeam Dose Engine, a product of Neutron Therapeutics (Finland) The nuBeam Dose Engine is a Monte Carlo dose calculation software package designed by Neutron Therapeutics in Helsinki, Finland to provide NCT dose calculation functionality specifically for use with RayStation and nuBeam. It is based on the open source Geant4 Monte Carlo simulation toolkit. The nuBeam Dose Engine is also part of the clinical investigation and is considered safe and effective based on in-phantom verification of the delivered dose.

Summary of relevant characteristics of nuBeam

The key features of the nuBeam Suite are:

* A therapeutically useful neutron beam intensity for NCT with a flux >109 n/cm2/s at the output plane.
* A neutron beam energy distribution tailored for NCT, primarily "epithermal neutrons": 0.5 eV < En < 10 keV.
* A well collimated and shielded beam aperture to appropriately confine the neutrons to the target region of the body.
* A robotically controlled patient positioning system for automated control of the patient position during irradiation.
* In-room CT imaging of the patient for image guided radiation therapy
* Precise on-line monitoring of the neutron beam to ensure the prescribed number of monitor units are delivered to the patient.
* Comprehensive NCT planning capability to accurately calculate the neutron flux distribution within the patient and thereby estimate the radiation dose delivered by the system.

Indications for Use

Neutron Therapeutics proposes the following draft of the indication for use statement:

"The nuBeam Suite is a medical device designed to produce and deliver a neutron beam for the treatment of patients with localized tumors and other conditions susceptible to treatment by Boron Neutron Capture Therapy (BNCT)."

nuBeam Therapeutic Neutron Source

The nuBeam Therapeutic Neutron Source (TNS) is the primary investigational device in this clinical study. It is composed of three major subsystems:

1. The Neutron Source System (NSS)
2. The On-Line Beam Monitoring System (OLBMS)
3. Treatment Control System (TCS) The Neutron Source System (NSS) is an accelerator-based system comprising an electrostatic proton accelerator, a rotating solid lithium neutron generating target, and a neutron beam shaping assembly to deliver the clinical neutron beam. The On-Line Beam Monitoring System (OLBMS) monitors the neutron fluence delivered to the patient to match the plan. The Treatment Control System (TCS) controls the operation of the nuBeam Suite during patient setup and radiation delivery.

The Neutron Source System (NSS) produces a neutron beam with key attributes similar to the FiR-1 reactor-based neutron source that was previously used to administer NCT in Finland. These beam attributes include the high epithermal neutron flux, low fast neutron dose level, low thermal neutron dose level, and low gamma dose level. A plot of the comparison between the FiR-1 and nuBeam neutron spectra. Beam delimiter materials and sizes are identical to the FiR-1 system. Because of this similarity in output, it is possible to build on the clinical evidence that has already been obtained at FiR-1.

Helsinki University Hospital has received a license to use the system from the STUK (Finnish nuclear and radiation safety authority) prior to use in the clinical investigation. The license is granted in two phases:

* License to operate the system for testing purposes (Licensing Phase I, completed)
* License to operate the system for clinical purposes (Licensing Phase II, to be applied during the trial process)

Granting of the phase I license indicates that the STUK is satisfied with the shielding and radiation safety measures that Helsinki University Hospital and Neutron Therapeutics have undertaken in the design and implementation of the facility. Granting of the phase II license indicates that the STUK is satisfied with the patient safety considerations and hazard mitigation measures undertaken by Helsinki University Hospital and Neutron Therapeutics.

Manufacturing and any special handling

The major components of the nuBeam Suite are assembled by the manufacturers at their respective manufacturing sites and tested against subsystem level requirements prior to shipment to the customer (Helsinki University Hospital) site. Once fully assembled at the customer site, all system level tests and calibrations are performed.

The main component of the system, the TNS, is assembled first at the Neutron Therapeutics manufacturing site in Danvers, Massachusetts, USA and tested prior to shipment at full proton beam output and low intensity neutron output.

Full neutron output operation is only conducted at the customer site due to shielding and neutron activation restrictions.

The system is a fixed installation device in a controlled access indoor climate-controlled environment. During operation, certain materials become radioactive. Requirements for the handling of radioactive materials during service and maintenance will follow STUK radiation authority guidelines and the instructions contained in the nuBeam service manuals.

Labeling and Instructions for Use (IFU)

The investigational devices are clearly labeled as an investigational device. The basic steps for using the nuBeam Suite to deliver an NCT irradiation are as follows:

1. Therapeutic Neutron Source preparation/calibration
2. CT imaging of the target region
3. Position of the patient
4. Irradiation to the planned dose
5. Close-out/Shutdown A copy of the Instructions for Use / User Guide(s) will be provided within the nuBeam Suite. The device must always be used according to the Instructions for Use.

nuBeam users and service personnel are made aware of potentially hazardous situations that have been identified in the Risk Management process, through operator training and the use of labeling consisting of User Guides and physically applied labels and signage. The use of internationally recognized symbology describing hazards are employed when applicable. The primary hazards identified for which the user is made aware include: radiation, electric shock, electromagnetic, thermal, functional and use error.

For radiation hazards, STUK labeling guidelines were applied (ST 1.3, Warnings for Radiation Sources).

The potential risks, warnings, precautions, and contra-indications associated with the use of the device are described further in the Investigator Brochure and in Section 11 Benefits and Risks.

Mechanism of action of boron neutron capture therapy BNCT is a biologically targeted form of radiation therapy. It is a binary therapy, meaning it relies on the interaction between an applied radiation field and an administered pharmaceutical. The patient first receives an intravenous infusion of a drug containing the isotope boron-10 (a 'boron carrier'). This drug is designed to cause the boron-10 to preferentially accumulate in tumor cells with a concentration that is higher than that in healthy tissues. A typical goal for the ratio of boron in cancer to healthy tissue is 3:1 or higher. When the target area is then exposed to thermal neutrons, they are absorbed by boron-10. This neutron capture reaction leads to the emission of high-energy charged particles: alpha particles and Li-7 (lithium-7) recoil nuclei. These particles have short range (<10 μm, roughly the diameter of a cell). The charged particles comprise the therapeutic radiation and are created preferentially in cells with high boron-10 concentration. Hence BNCT can in principle target cancerous tissue at the cellular level, while sparing healthy tissue. A certain concentration of boron-10 is necessary to achieve a 'boron dose' that is much higher than the dose delivered by the neutron beam itself. A typical goal for the boron-10 concentration in cancer cells is ≥20 μg/g.

The alpha particles and Li-7 reaction products also have the property of "high linear energy transfer" (high LET) meaning a large amount of energy is deposited over a short path length. High LET radiation causes extensive DNA damage that is often unrepairable and leads directly to cell death. Hence why BNCT has the potential for greater success to reduce or eliminate tumors. For conventional radiation therapy, fractionation is used to take advantage of healthy tissue's generally enhanced ability to repair the damage compared to cancerous tissue. For the high-LET radiation in BNCT there is not expected to be any benefit to fractionation.

INVESTIGATIONAL DRUG/MEDICINAL PRODUCT

L-boronophenylalanine (L-BPA) will be purchased from a commercial source. The manufacturer is Interpharma Praha in Prague, Czech, and L-BPA is imported into Finland by pharmaceutical wholesaler Tamro. HUH hospital pharmacy and Tamro performed a joint Good Manufacturing Practice (GMP) audit to the manufacturer in 15.2.2018 and found no critical deficiencies in the production and QC of L-BPA.

In the current trial the dose of L-BPA administered will be 400 mg per kilogram of the body weight, complexed with fructose to increase solubility. This L-BPA dose was selected based on a Phase I dose escalation trial carried out in an adult patient population with histologically confirmed malignant glioma that had progressed after surgery and external beam radiotherapy, In this dose escalation study, the 400 mg/kg L-BPA dose infused over 2 hours prior to neutron irradiation was found optimal compared to the other dose levels evaluated (290 mg/kg, 350 mg/kg, and 450 mg/kg) in the glioma patient population. Subsequently, the 400 mg/kg dose was selected to be used in a clinical trial where patients with locally recurred, inoperable head and neck cancer were treated with BNCT. The 400 mg/kg dose was well tolerated in a patient population with head and neck cancer, and most the study patients achieved objective response to L-BPA-mediated BNCT. Therefore, the L-BPA dose of 400 mg/kg, administered complexed with fructose over 2 hours prior to neutron irradiation, was selected for the current trial.

Hospital pharmacy will compound the L-BPA with fructose to create L-BPA 30 g/L fructose complex solution for infusion, as pure L-BPA has low solubility, and it is irritating during infusion. The complex is created by weighing L-BPA and fructose, adding water, raising the pH of the solution to ≈10, and heating and stirring of the solution. Finally, the pH is adjusted to 7,6 and the solution is stored overnight to maximize the complexation. Next day the solution is sterile filtered in a GMP class A laminar flow cabinet and packaged to an infusion bottle or infusion bag. During filtration quality control (QC) samples are taken and endotoxins are tested with a chromokinetic quick test (acceptance limit 175 EU/V). Finally, the infusion package is labeled and delivered to the Comprehensive Cancer Center. The shelf-life of the infusion is 24 hours as calculated from the end of sterile filtration.

Each study subject dose is prepared individually ex tempore, based on the study subject weight provided by the principal investigator or study nurse. Production and QC is documented by the hospital pharmacy and a qualified pharmaceutical person releases the dose based on the documentation. Hospital pharmacy maintains a log of all manufactured doses.

STUDY OBJECTIVES, DESIGN, AND OUTCOMES This is an open-label, 1-group, prospective, non-randomized, single-center, Phase I study. The study objective is to evaluate the safety and efficacy of BNCT using the nuBeam Suite as a trial treatment of locally and/or locoregionally recurrent, inoperable head and neck carcinoma previously irradiated with conventional radiotherapy.

The study has a radiation dose escalation design, consisting of three cohorts of 3, 3, and 4 study subjects for 10 study subjects in total to demonstrate safety. A new cohort can be initiated when the last study subject of the previous cohort has been followed up for at least 3 weeks. If no acute toxicity greater than 3 is detected, the next cohort of study subjects will be treated.

Objective(s)/Endpoints:

Primary Endpoint The primary objective is to assess the safety of accelerator-based neutron radiation using the nuBeam Suite, and explicitly, the nuBeam Treatment Delivery System (TDS) in delivering BNCT to treat cancer patients. Safety/toxicity of neutron radiation delivered by the nuBeam TDS will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 at one month after the last BNCT trial treatment.

Secondary Endpoints

Secondary Performance/Efficacy Endpoint:

* Trial Irradiation Success for the nuBeam TDS: defined as the ability to deliver the planned radiation dose to the target site at each BNCT trial treatment.
* Procedure success of the nuBeam Suite: defined as the ability to plan the trial treatment using the trial treatment planning software, position and target the tumor site using the robotic table in conjunction with the CT scanner and calculate the required radiation dose for each planned BNCT trial treatment.
* Treatment effectiveness:

  * to assess the response rate of locally and/or locoregionally recurrent, inoperable head and neck carcinoma previously irradiated with conventional radiotherapy to BNCT. The responses will be assessed periodically until 24 months since the second BNCT according to RECIST 1.v1, and the best response achieved will be recorded.

In addition to the objective response rate (ORR), the following parameters will be assessed:

* Duration of response to BNCT
* The clinical benefit rate (CBR) - includes complete response, partial response, and stabilized disease for a minimum of 8 weeks since the date of the first BNCT.
* Locoregional recurrence-free survival (LRFS)
* Progression-free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

1. The patient considered for the study has provided a written informed consent as approved by the EC prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. ≥ 18 years of age at the time of enrollment.
3. Histologically confirmed head and neck carcinoma.
4. Inoperable cancer, prior surgery may or may not have been done.
5. Prior radiotherapy or chemoradiotherapy has been given.
6. Anticipated life expectancy of at least 6 months.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

1. Presence of distant metastases.
2. World Health Organization (WHO) performance status > 2 (see Appendix 2).
3. Concurrent uncontrolled localized cancer other than head and neck carcinoma or overtly metastatic cancer.
4. The patient has access to a non-experimental, effective treatment option and is a suitable candidate for such therapy.
5. Concomitant chemotherapy.
6. Concurrent experimental therapy or participation in a trial with an experimental therapy within 3 months prior to study inclusion.
7. Less than 3 months since prior radiation therapy.
8. Major surgery within 4 weeks prior to study inclusion.
9. Unremovable metal implants present in the head and neck region that will interfere with CT/MRI-based dose-planning.
10. Known sensitivity to the study drug.
11. One or more of the following:

    * Blood hemoglobin < 100 g/L, neutrophils < 1.5 x 109/L, platelet count < 120 x 109/L
    * Serum/plasma creatinine > 1.5 x Upper Limit of Normal (ULN)
    * Serum bilirubin 2.0 > ULN
    * Serum ALT and/or AST > 2.0 x ULN
    * Serum alkaline phosphatase > 2.5 x ULN
12. Serious uncontrolled infection or other serious uncontrolled concomitant disease.
13. Collagen vascular disease or a disease that is considered to increase radiosensitivity of normal tissues to radiation (e.g., ataxia-telangiectasia)
14. The patient is unwilling or unable to comply with the CIP required follow-up visits for the duration of the study.
15. Untreated or severe treated congestive heart failure, cardiac pacemaker, or renal failure.
16. Restlessness or inability to lie in a cast for about 30 minutes.
17. Clinical follow-up after therapy cannot be arranged or the patient is not willing to participate in the follow-up.
18. Known pregnancy, breastfeeding, or planning of pregnancy; for women of childbearing potential, a negative urine pregnancy test must be obtained prior to enrollment.
19. The patient is not able to understand the nature of the study and trial treatment options.
20. Phenylketonuria.
21. Fructose intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | The expected duration to the primary outcome is 13 months. The primary safety endpoint is 1 month after the final/2nd BNCT trial treatment of the last study subject. Study subject enrollment is anticipated to take 12 months.
  The primary objective is to assess the safety of accelerator-based neutron radiation using the nuBeam Suite, and explicitly, the nuBeam Treatment Delivery System (TDS) in delivering BNCT to treat cancer patients. Safety/toxicity of neutron radiation delivered by the nuBeam TDS will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 at one month after the last BNCT trial treatment.

SECONDARY OUTCOMES:
Trial Irradiation Success for the nuBeam TDS | The expected duration to the primary outcome is 13 months. The primary safety endpoint is 1 month after the final/2nd BNCT trial treatment of the last study subject. Study subject enrollment is anticipated to take 12 months.
  Ability to deliver the planned radiation dose to the target site at each BNCT trial treatment.
Procedure success of the nuBeam Suite | The expected duration to the primary outcome is 13 months. The primary safety endpoint is 1 month after the final/2nd BNCT trial treatment of the last study subject. Study subject enrollment is anticipated to take 12 months.
  Ability to plan the trial treatment using the trial treatment planning software, position and target the tumor site using the robotic table in conjunction with the CT scanner and calculate the required radiation dose for each planned BNCT trial treatment.
Treatment effectiveness | The expected duration to the primary outcome is 13 months. The primary safety endpoint is 1 month after the final/2nd BNCT trial treatment of the last study subject. Study subject enrollment is anticipated to take 12 months.
  Assess the overall response rate (ORR) of locally and/or locoregionally recurrent, inoperable head and neck carcinoma previously irradiated with conventional radiotherapy to BNCT. The responses will be assessed periodically until 24 months since the second BNCT according to RECIST 1.v1, and the best response achieved will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Estrada, PhD, Study Chair — Neutron Therapeutics
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Not yet decided

REFERENCES:
- [Background] Salama JK, Vokes EE, Chmura SJ, Milano MT, Kao J, Stenson KM, Witt ME, Haraf DJ. Long-term outcome of concurrent chemotherapy and reirradiation for recurrent and second primary head-and-neck squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):382-91. doi: 10.1016/j.ijrobp.2005.07.005. Epub 2005 Oct 5. PMID 16213104
- [Background] Igaki H, Murakami N, Nakamura S, Yamazaki N, Kashihara T, Takahashi A, Namikawa K, Takemori M, Okamoto H, Iijima K, Chiba T, Nakayama H, Takahashi A, Kaneda T, Takahashi K, Inaba K, Okuma K, Nakayama Y, Shimada K, Nakagama H, Itami J. Scalp angiosarcoma treated with linear accelerator-based boron neutron capture therapy: A report of two patients. Clin Transl Radiat Oncol. 2022 Feb 18;33:128-133. doi: 10.1016/j.ctro.2022.02.006. eCollection 2022 Mar. PMID 35252597
- [Background] Bokstein F, Blumenthal DT, Corn BW, Gez E, Matceyevsky D, Shtraus N, Ram Z, Kanner AA. Stereotactic radiosurgery (SRS) in high-grade glioma: judicious selection of small target volumes improves results. J Neurooncol. 2016 Feb;126(3):551-7. doi: 10.1007/s11060-015-1997-5. Epub 2015 Nov 24. PMID 26603164
- [Background] Kawabata S, Suzuki M, Hirose K, Tanaka H, Kato T, Goto H, Narita Y, Miyatake SI. Accelerator-based BNCT for patients with recurrent glioblastoma: a multicenter phase II study. Neurooncol Adv. 2021 May 20;3(1):vdab067. doi: 10.1093/noajnl/vdab067. eCollection 2021 Jan-Dec. PMID 34151269
- [Background] Hirose K, Konno A, Hiratsuka J, Yoshimoto S, Kato T, Ono K, Otsuki N, Hatazawa J, Tanaka H, Takayama K, Wada H, Suzuki M, Sato M, Yamaguchi H, Seto I, Ueki Y, Iketani S, Imai S, Nakamura T, Ono T, Endo H, Azami Y, Kikuchi Y, Murakami M, Takai Y. Boron neutron capture therapy using cyclotron-based epithermal neutron source and borofalan (10B) for recurrent or locally advanced head and neck cancer (JHN002): An open-label phase II trial. Radiother Oncol. 2021 Feb;155:182-187. doi: 10.1016/j.radonc.2020.11.001. Epub 2020 Nov 11. PMID 33186684
- [Background] Barth RF, Zhang Z, Liu T. A realistic appraisal of boron neutron capture therapy as a cancer treatment modality. Cancer Commun (Lond). 2018 Jun 19;38(1):36. doi: 10.1186/s40880-018-0280-5. PMID 29914575
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] H, Järvinen and W. Voorbraak (eds.),Recommendations for the Dosimetry of Boron Neutron Capture Therapy, NRG Report 21425/03.55339/C, Petten, The Netherlands, 2003
- [Background] Kawabata S, Hiramatsu R, Kuroiwa T, Ono K, Miyatake S. Boron neutron capture therapy for recurrent high-grade meningiomas. J Neurosurg. 2013 Oct;119(4):837-44. doi: 10.3171/2013.5.JNS122204. Epub 2013 Jun 28. PMID 23808536
- [Background] Menendez PR, Roth BM, Pereira MD, Casal MR, Gonzalez SJ, Feld DB, Santa Cruz GA, Kessler J, Longhino J, Blaumann H, Jimenez Rebagliati R, Calzetta Larrieu OA, Fernandez C, Nievas SI, Liberman SJ. BNCT for skin melanoma in extremities: updated Argentine clinical results. Appl Radiat Isot. 2009 Jul;67(7-8 Suppl):S50-3. doi: 10.1016/j.apradiso.2009.03.020. Epub 2009 Mar 27. PMID 19375342
- [Background] Wang LW, Chen YW, Ho CY, Hsueh Liu YW, Chou FI, Liu YH, Liu HM, Peir JJ, Jiang SH, Chang CW, Liu CS, Lin KH, Wang SJ, Chu PY, Lo WL, Kao SY, Yen SH. Fractionated Boron Neutron Capture Therapy in Locally Recurrent Head and Neck Cancer: A Prospective Phase I/II Trial. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):396-403. doi: 10.1016/j.ijrobp.2016.02.028. Epub 2016 Feb 13. PMID 27084657
- [Background] Suzuki M, Kato I, Aihara T, Hiratsuka J, Yoshimura K, Niimi M, Kimura Y, Ariyoshi Y, Haginomori S, Sakurai Y, Kinashi Y, Masunaga S, Fukushima M, Ono K, Maruhashi A. Boron neutron capture therapy outcomes for advanced or recurrent head and neck cancer. J Radiat Res. 2014 Jan 1;55(1):146-53. doi: 10.1093/jrr/rrt098. Epub 2013 Aug 16. PMID 23955053
- [Background] Aihara T, Morita N, Kamitani N, Kumada H, Ono K, Hiratsuka J, Harada T. BNCT for advanced or recurrent head and neck cancer. Appl Radiat Isot. 2014 Jun;88:12-5. doi: 10.1016/j.apradiso.2014.04.007. Epub 2014 Apr 21. PMID 24799334
- [Background] Kato I, Fujita Y, Maruhashi A, Kumada H, Ohmae M, Kirihata M, Imahori Y, Suzuki M, Sakrai Y, Sumi T, Iwai S, Nakazawa M, Murata I, Miyamaru H, Ono K. Effectiveness of boron neutron capture therapy for recurrent head and neck malignancies. Appl Radiat Isot. 2009 Jul;67(7-8 Suppl):S37-42. doi: 10.1016/j.apradiso.2009.03.103. Epub 2009 Apr 2. PMID 19409799
- [Background] Kankaanranta L, Seppala T, Koivunoro H, Saarilahti K, Atula T, Collan J, Salli E, Kortesniemi M, Uusi-Simola J, Valimaki P, Makitie A, Seppanen M, Minn H, Revitzer H, Kouri M, Kotiluoto P, Seren T, Auterinen I, Savolainen S, Joensuu H. Boron neutron capture therapy in the treatment of locally recurred head-and-neck cancer: final analysis of a phase I/II trial. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e67-75. doi: 10.1016/j.ijrobp.2010.09.057. Epub 2011 Feb 6. PMID 21300462
- [Background] Kankaanranta L, Seppala T, Koivunoro H, Saarilahti K, Atula T, Collan J, Salli E, Kortesniemi M, Uusi-Simola J, Makitie A, Seppanen M, Minn H, Kotiluoto P, Auterinen I, Savolainen S, Kouri M, Joensuu H. Boron neutron capture therapy in the treatment of locally recurred head and neck cancer. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):475-82. doi: 10.1016/j.ijrobp.2007.03.039. Epub 2007 Aug 6. PMID 17689034
- [Background] Barth RF, Vicente MG, Harling OK, Kiger WS 3rd, Riley KJ, Binns PJ, Wagner FM, Suzuki M, Aihara T, Kato I, Kawabata S. Current status of boron neutron capture therapy of high grade gliomas and recurrent head and neck cancer. Radiat Oncol. 2012 Aug 29;7:146. doi: 10.1186/1748-717X-7-146. PMID 22929110
- [Background] Kim YS. Reirradiation of head and neck cancer in the era of intensity-modulated radiotherapy: patient selection, practical aspects, and current evidence. Radiat Oncol J. 2017 Mar;35(1):1-15. doi: 10.3857/roj.2017.00122. Epub 2017 Mar 31. PMID 28395502
- [Background] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Background] Argiris A, Li Y, Forastiere A. Prognostic factors and long-term survivorship in patients with recurrent or metastatic carcinoma of the head and neck. Cancer. 2004 Nov 15;101(10):2222-9. doi: 10.1002/cncr.20640. PMID 15452834
- [Background] De Felice F, Polimeni A, Valentini V, Brugnoletti O, Cassoni A, Greco A, de Vincentiis M, Tombolini V. Radiotherapy Controversies and Prospective in Head and Neck Cancer: A Literature-Based Critical Review. Neoplasia. 2018 Mar;20(3):227-232. doi: 10.1016/j.neo.2018.01.002. Epub 2018 Feb 12. PMID 29448084
- [Background] Peng G, Wang T, Yang KY, Zhang S, Zhang T, Li Q, Han J, Wu G. A prospective, randomized study comparing outcomes and toxicities of intensity-modulated radiotherapy vs. conventional two-dimensional radiotherapy for the treatment of nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):286-93. doi: 10.1016/j.radonc.2012.08.013. Epub 2012 Sep 17. PMID 22995588
- [Background] Nutting CM, Morden JP, Harrington KJ, Urbano TG, Bhide SA, Clark C, Miles EA, Miah AB, Newbold K, Tanay M, Adab F, Jefferies SJ, Scrase C, Yap BK, A'Hern RP, Sydenham MA, Emson M, Hall E; PARSPORT trial management group. Parotid-sparing intensity modulated versus conventional radiotherapy in head and neck cancer (PARSPORT): a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2011 Feb;12(2):127-36. doi: 10.1016/S1470-2045(10)70290-4. Epub 2011 Jan 12. PMID 21236730
- [Background] Marur S, Forastiere AA. Head and Neck Squamous Cell Carcinoma: Update on Epidemiology, Diagnosis, and Treatment. Mayo Clin Proc. 2016 Mar;91(3):386-96. doi: 10.1016/j.mayocp.2015.12.017. PMID 26944243
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103